CLINICAL TRIAL: NCT05820191
Title: B-amyloid as a Marker for GBM Bioimaging
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Central del Caribe (Other)
Collaborators: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Lilia Kucheryavykh, Associate Professor, Universidad Central del Caribe
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMY-GBM
Record Dates: First submitted 2023-03-13; First posted 2023-04-19 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Glioblastoma
Keywords: Glioblastoma, Amyvid
MeSH Terms: conditions — Glioblastoma | interventions — florbetapir

STUDY DESIGN:
Intervention Model Description: 3 patients, diagnosed with GBM, who underwent tumor resection surgery with concurrent chemo- and/or radiotherapy and developed enlarging tumor lesion, will be involved to the study. PET-CT with use of Amyvid radioisotope tracer will be performed for 3 study participants. Amyvid-PET images will be analyzed together with previously performed MRI, MRS and MRP images, to identify pattern of deposition in tumor and peri-tumoral areas of brain.Tissue specimens, separated from total tumor after planned surgical resection and prior Amyvid-PET analysis, will be analyzed to identify amyloid-β expression level, tumor phenotype and vascularization. Data will be correlated with PET images to determine whether Amyvid-positive patterns represent distinct tumor phenotype.
Masking Description: Double blinding analysis of PET images will be performed. Involved Radiologists will provide their independent opinions. In addition, blinding research strategy with withholding of patient information, with three independent people involved for data collection and analysis will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AMY-GBM (Experimental): Amyvid-PET scan will be performed. According to approved protocol for Alzheimer's disease diagnostics, 370MBq (10mCi) absorbed dose 7mSv of Amyvid will be introduced intravenously and 30-50 minutes after the PET images will be acquired.
  Interventions: Drug: Amyvid, Intravenous Solution

INTERVENTIONS:
Drug: Amyvid, Intravenous Solution — Amyvid 370MBq (10mCi) absorbed dose 7mSv of will be introduced intravenously and 30-50 minutes after the PET images will be acquired.
  Other Names: Florbetapir-f18

SUMMARY:
This project is aimed at improvement of glioblastoma (GBM) diagnostic strategies for discrimination of tumor progression and chemo- and radiotherapeutic treatment-related changes in brain tissue. The study will elucidate the diagnostic value of PET imaging with use of amyloid-β radioisotope tracer Amyvid (Florbetapir F18) for GBM. The results of the study will provide data for development of new approach for GBM diagnostics.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is one of the most malignant forms of brain cancer. Majority of GBMs relapse shortly after tumor resection, and the timely follow-up diagnosis and treatment is vital for patient's survival. However, chemo- and radiotherapeutic treatment of GBM patients cause metabolic and structural changes in brain parenchyma, manifested as metabolic and matrix remodeling modifications, and mimic tumor progression in magnetic resonance imaging (MRI) images. This creates difficulties in discrimination of real tumor progression and post-treatment modifications. No current imaging techniques, including MRI, magnetic resonance spectroscopy (MRS) or perfusion MR (MRP) can provide effective determination of tumor progression and treatment-related changes of brain tissue, that represents current unmet clinical need. The goal of the study is to identify specific biomarker for GBM, that can be used for precise imaging and diagnostics.

The accumulation of amyloid-β in human GBM specimens and in mouse glioma implantation model was previously demonstrated. Intravenous administration of amyloid-β marker thioflavin T resulted in accumulation of fluorescence in brain tumors in mouse GBM model 15 minutes after administration and allowed detailed visualization of tumor structure with use of confocal microscopy. The hypothesis of the study is that Amyvid (Florbetapir F18), a radioisotope tracer, that binds amyloid aggregates and is currently used for brain PET diagnostics of Alzheimer disease, can be used as a safe and effective marker for PET diagnostics of recurrent GBM.

The central study question: if Amyvid-PET provides visualization of GBM tumors and discriminate recurrent tumor and post-treatment tissue modifications in human brain, and thus presents the potential for amyloid-binding radioisotope tracers as GBM diagnostic tool. The purpose of the study is to characterize and describe the ability of Amyvid to reach GBM tumor in humans and to bind specific tumor structures as necrotic, middle and invasion areas of tumor, as well as blood vessel structures and extracellular matrix in tumor. The study is designed as human clinical trials phase 2A.

ELIGIBILITY:
Inclusion Criteria:

* GBM diagnose confirmed by MRI and histopathology
* Had undergone gross total or subtotal resection of their tumor and developed enlarging and/or new enhancing lesion(s), recommended for second resection
* Had or had not received radiation therapy with concomitant and adjuvant TMZ chemotherapy
* Had pre-operative and follow up conventional MRI, MRS and/or Perfusion MR scans, available for analysis

Exclusion Criteria:

• Previous allergic reaction to radioisotope tracers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of Amyvid deposition in GBM tumor structures | Through study completion, an average of 1 year
  The Amyvid patterns of deposition (brightness or darkness patterns) will be analyzed in whole brain, tumor and peri-tumor resection region with and without representation of post-treatment modifications, as compared to MRI scans.
Correlation of Amyvid deposition with components of high metabolic activity. | Through study completion, an average of 1 year
  Association of Amyvid deposition patterns with brain tissue components of high and low metabolic activity will be analyzed as compared to MRS images.
Correlation of Amyvid deposition with components of increased vascularization. | Through study completion, an average of 1 year
  Association of Amyvid deposition patterns with areas of high and low vascularization will be analyzed as compared to MRP scans.

SECONDARY OUTCOMES:
Correlation of Amyvid deposition and amyloid- β expression in GBM specimens. | Through study completion, an average of 1 year
  Tissue specimens, separated from total tumor after planned surgical resection and prior Amyvid-PET analysis, will be analyzed by western blot to quantify amyloid-β expression level and correlate with deposition of Amyvid, as identified by Amyvid-PET.
Correlation of Amyvid deposition with characteristics of tumor vasculature in GBM specimens. | Through study completion, an average of 1 year
  Tissue specimens, separated from total tumor after planned surgical resection and prior Amyvid-PET analysis, will be analyzed with use of immunofluorescence imaging of blood vessels to characterize tumor vasculature structure (as capillary density and diameter) and correlate with deposition of Amyvid, as identified by Amyvid-PET.

CONTACTS AND LOCATIONS:
Overall Officials: Lilia Kucheryavykh, PhD, Principal Investigator — Universidad Central del Caribe (Central University of the Caribbean)
Locations (2):
- Puerto Rico (2):
  - Central University of the Caribbean (UCC), Bayamón, PR
  - University of Puerto Rico, Medical Science Campus, San Juan

IPD SHARING:
Plan to Share IPD: No
Investigation will be performed on anonymous basis in order to protect the confidentiality of the subjects.

REFERENCES:
- [Background] Kucheryavykh LY, Ortiz-Rivera J, Kucheryavykh YV, Zayas-Santiago A, Diaz-Garcia A, Inyushin MY. Accumulation of Innate Amyloid Beta Peptide in Glioblastoma Tumors. Int J Mol Sci. 2019 May 20;20(10):2482. doi: 10.3390/ijms20102482. PMID 31137462
- [Background] Zayas-Santiago A, Diaz-Garcia A, Nunez-Rodriguez R, Inyushin M. Accumulation of amyloid beta in human glioblastomas. Clin Exp Immunol. 2020 Dec;202(3):325-334. doi: 10.1111/cei.13493. Epub 2020 Aug 11. PMID 32654112
- [Background] Kucheryavykh LY, Davila-Rodriguez J, Rivera-Aponte DE, Zueva LV, Washington AV, Sanabria P, Inyushin MY. Platelets are responsible for the accumulation of beta-amyloid in blood clots inside and around blood vessels in mouse brain after thrombosis. Brain Res Bull. 2017 Jan;128:98-105. doi: 10.1016/j.brainresbull.2016.11.008. Epub 2016 Nov 28. PMID 27908798